CLINICAL TRIAL: NCT01881126
Title: An Efficacy and Safety Study of Bimatoprost 0.01% Alone Compared With Travoprost 0.004% and Timolol 0.5% in Subjects With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMA-LUM-12-021
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Travoprost; Timolol; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimatoprost 0.01% and hypromellose 0.3% (Active Comparator): Bimatoprost 0.01% and hypromellose 0.3% lubricant eye drops (for masking purposes) each administered to both eyes once daily for 12 weeks.
  Interventions: Drug: bimatoprost 0.01%; Drug: hypromellose 0.3%
- travatan 0.004% and timolol 0.5% (Active Comparator): Travatan 0.004% and timolol 0.5% each administered to both eyes once daily for 12 weeks.
  Interventions: Drug: travatan 0.004%; Drug: timolol 0.5%

INTERVENTIONS:
Drug: bimatoprost 0.01% — Bimatoprost 0.01% administered to both eyes once daily for 12 weeks.
  Other Names: Lumigan® RC; Lumigan®
  Arms: bimatoprost 0.01% and hypromellose 0.3%
Drug: travatan 0.004% — Travatan 0.004% administered to both eyes once daily for 12 weeks.
  Other Names: Travatan Z®
  Arms: travatan 0.004% and timolol 0.5%
Drug: timolol 0.5% — Timolol 0.5% administered to both eyes once daily for 12 weeks.
  Other Names: Timolol Maleate-EX; Timolol GFS
  Arms: travatan 0.004% and timolol 0.5%
Drug: hypromellose 0.3% — Hypromellose 0.3% lubricant eye drops (for masking purposes) administered to both eyes once daily for 12 weeks.
  Other Names: GenTeal®
  Arms: bimatoprost 0.01% and hypromellose 0.3%

SUMMARY:
This efficacy and safety study will evaluate LUMIGAN® RC/ LUMIGAN® .01 (bimatoprost 0.01%) alone compared to TRAVATAN Z® (travoprost 0.004%) and TIMOLOL MALEATE-EX, 0.5%/TIMOLOL GFS 0.5% (timolol 0.5% ophthalmic gel forming solution) in patients who require IOP lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or glaucoma that requires treatment with medication
* Have a best corrected visual acuity (BCVA) of 20/100 or better in both eyes

Exclusion Criteria:

* History of LASIK, LASEK, RK, and/or PRK in the study eye(s)
* History of any intraocular surgery or glaucoma laser surgery in the study eye(s) within 3 months
* Use of topical, periorbital, intravitreal or systemic steroid within 3 months or expected use during the course of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Canada (2):
  - Barrie, Ontario
  - Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.01% and Hypromellose 0.3% | Travatan 0.004% and Timolol 0.5%
Started | 47 | 46
Completed | 46 | 44
Not Completed | 1 | 2
Not completed — Non-compliance | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.01% and Hypromellose 0.3% | Travatan 0.004% and Timolol 0.5% | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (9.34) | 67.3 (8.19) | 67.5 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 23 | 28 | 51

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) in the Study Eye at 8 AM, 12 PM, and 4 PM
Description: IOP is a measurement of the fluid pressure inside the eye. IOP of the study eye (worse eye) is measured at 8 AM, 12 PM, and 4 PM. IOP is either the average of 2 measurements, or, if a third measurement is required, the average of 3 measurements.
Time Frame: Week 12 at 8 AM, 12 PM, and 4 PM
Population: Intent-to-Treat: all subjects who were randomized to study medication
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.01% and Hypromellose 0.3% | Travatan 0.004% and Timolol 0.5%
Number analyzed (Participants) | 46 | 44
Millimeters of Mercury (mmHg)
  Week 12 at 8 AM | 16.4 (0.46) | 15.1 (0.43)
  Week 12 at 12 PM | 16.0 (0.49) | 15.0 (0.38)
  Week 12 at 4 PM | 16.5 (0.48) | 14.5 (0.34)

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.01% and Hypromellose 0.3% | Travatan 0.004% and Timolol 0.5%
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/46
Other Adverse Events (participants affected / at risk) | 0/47 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.01% and Hypromellose 0.3% (N=47) | Travatan 0.004% and Timolol 0.5% (N=46)
Angina Pain (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.